CLINICAL TRIAL: NCT01856387
Title: the Predictive Value of neutrophil-to Lymphocyte Ratio on Preeclampsia- Eclampsia
Brief Title: The Effect of neutrophil-to Lymphocyte Ratio in Preeclampsia- Eclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Ayse Kirbas, Ayse Kirbas, MD, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: Zekai Tahir Burak
Record Dates: First submitted 2013-05-04; First posted 2013-05-17 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2013-05

CONDITIONS: Preeclampsia; Eclampsia
Keywords: preeclampsia; eclampsia; prediction; neutrophil-to Lymphocyte ratio
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — whole blood, serum, white cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normal pregnancy outcomes: do not expect poor pregnancy outcomes on normal patients
  Interventions: Biological: high neutrophil to lymphocyte ratio; Other: normal neutrophil-to Lymphocyte ratio
- adverse pregnancy outcome: high ratio of Neutrophil / lymphocyte ratio may predict preeclampsia eclampsia
  Interventions: Biological: high neutrophil to lymphocyte ratio; Other: normal neutrophil-to Lymphocyte ratio

INTERVENTIONS:
Biological: high neutrophil to lymphocyte ratio
Other: normal neutrophil-to Lymphocyte ratio

SUMMARY:
Neutrophil/lymphocyte ratio (NLR) is a marker of systemic inflammation and endothelial dysfunction. In recent years, it has been reported that the individual components of the differential white cell count, specifically the neutrophil and lymphocyte counts,may have clinical utility in predicting diseases. An elevated NLR has been shown to be a prognostic indicator in various malignancies. İn the literature, many studies have been shown that NLR have predictive value in determining the prognosis of various diseases (cardiac or noncardiac diseases ). However, little is known about the predictive values of NLR in pregnancy complications. This study aimed to evaluate the potential predictive value of NLR in preeclampsia- eclampsia.

DETAILED DESCRIPTION:
In recent years, have been reported that the individual components of the differential white cell count, specifically the neutrophil and lymphocyte counts, may have clinical utility in predicting diseases.

An elevated NLR has been shown to be a prognostic indicator in various malignancies. İn the literatüre have been shown that NLR have predictive value in determining the prognosis of various diseases (cardiac or noncardiac diseases.However, little is known about the predictive values of NLR and PLR in gestational DM, preeclampsia and the other pregnancy complications.

Retrospective data were collected for patients who was diagnosed with , preeclampsia- eclampsia, The NLR was defined as the absolute neutrophil count divided by the absolute lymphocyte count.

ELIGIBILITY:
Inclusion Criteria:

pregnant women who developing preeclampsia eclampsia at pregnancy

Exclusion Criteria:

Known chronically maternal disease multiple pregnancy older than 40 years old

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: first trimester pregnant
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
the effect of neutrophil lymphocyte ratio in preeclampsia eclampsia | up to 6 months
  during 6 months ,the patients who was recorded with preeclampsi/eclampsia at our hospital ,first trimester whole blood count was taken and neutrophil lymphocyte ratio was calculated and recorded

CONTACTS AND LOCATIONS:
Overall Officials: ayse kirbas, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Turkey (Türkiye)